CLINICAL TRIAL: NCT04373031
Title: Induction Immunotherapy to Promote Immunologic Priming and Enhanced Response to Neoadjuvant Pembrolizumab + Chemotherapy in Triple Negative Breast Cancer (TNBC)
Brief Title: Pembrolizumab, IRX-2, and Chemotherapy in Triple Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Brooklyn ImmunoTherapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019000486
Record Dates: First submitted 2020-04-28; First posted 2020-05-04 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; IRX 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Control Arm: (Pembro + ACT): Pembrolizumab induction (single-dose 200mg IV), followed by pembrolizumab Q3W + paclitaxel (T) weekly x 4 cycles, followed by pembrolizumab + doxorubicin + cyclophosphamide (AC) Q3W x 4 cycles as neoadjuvant therapy prior to surgery.
  Interventions: Drug: Pembrolizumab
- Arm A (Experimental): • Arm A: (Pembro + IRX-2 + ACT): Pembrolizumab (single-dose 200mg IV) + cyclophosphamide (single-dose 300 mg/m2 IV) + IRX-2 induction (1mL SQ x 2 daily, x 10 days), followed by pembrolizumab Q3W + paclitaxel (T) weekly x 4 cycles, followed by IRX-2 re-induction (1mL SQ x 2 daily, x 10 days), followed by pembrolizumab + doxorubicin + cyclophosphamide (AC) Q3W x 4 cycles as neoadjuvant therapy prior to surgery.
  Interventions: Drug: Pembrolizumab; Drug: IRX 2

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a humanized anti-PD-1 mAb of the IgG4/kappa isotype with a stabilizing S228P sequence alteration in the Fc region.
  Other Names: KEYTRUDA
Drug: IRX 2 — IRX-2, is a cell-derived biologic with multiple active cytokine components that acts on multiple cell types of the immune system including T cells, dendritic cells and natural killer cells.
  Arms: Arm A

SUMMARY:
This is a Phase II, randomized, open-label trial to evaluate the clinical and immunologic activity of pembrolizumab plus chemotherapy when combined with various immunotherapy induction regimens as neoadjuvant therapy for triple negative breast cancer (TNBC).

DETAILED DESCRIPTION:
This is a Phase II, randomized, open-label trial to evaluate the clinical and immunologic activity of pembrolizumab plus chemotherapy when combined with various immunotherapy induction regimens as neoadjuvant therapy for triple negative breast cancer (TNBC).

A commonly used standard neoadjuvant regimen for TNBC is a weekly taxane (e.g., paclitaxel 80mg/m2) for 12 weeks followed by an anthracycline (e.g., doxorubicin 60 mg/m2 plus cyclophosphamide at 600 mg/m2 [AC]) every 3 weeks (Q3W) for 4 cycles.

The chemotherapy regimen included in this study is built upon the aforementioned regimen. Pembrolizumab in combination with this regimen will be studied as part of a multi-arm study that randomizes subjects to receive:

* Control Arm: (Pembro + ACT): Pembrolizumab induction (single-dose 200mg IV), followed by pembrolizumab Q3W + paclitaxel (T) weekly x 4 cycles, followed by pembrolizumab + doxorubicin + cyclophosphamide (AC) Q3W x 4 cycles as neoadjuvant therapy prior to surgery.
* Arm A: (Pembro + IRX-2 + ACT): Pembrolizumab (single-dose 200mg IV) + cyclophosphamide (single-dose 300 mg/m2 IV) + IRX-2 induction (1mL SQ x 2 daily, x 10 days), followed by pembrolizumab Q3W + paclitaxel (T) weekly x 4 cycles, followed by IRX-2 re-induction (1mL SQ x 2 daily, x 10 days), followed by pembrolizumab + doxorubicin + cyclophosphamide (AC) Q3W x 4 cycles as neoadjuvant therapy prior to surgery.
* Subsequent induction therapy arms are to be included in protocol amendments. Note: 1 cycle = 21 days

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial. The subject may also provide consent for Future Biomedical Research. However, the subject may participate in the main trial without participating in Future Biomedical Research.
2. Be a male or female subject greater than or equal to 18 years of age on day of signing informed consent.
3. Have locally confirmed TNBC, as defined by the most recent ASCO/CAP guidelines.
4. Have previously untreated locally advanced non-metastatic (M0) TNBC defined as the following combined primary tumor (T) and regional lymph node (N) staging per the current AJCC Version 8 staging criteria for breast cancer staging criteria as assessed by the investigator based on radiological and/or clinical assessment:

   * T1c, N1-N2
   * T2, N0-N2
   * T3, N0-N2
   * T4a-d, N0-N2 Note: bilateral tumors (i.e., synchronous cancers in both breasts) and/or multi-focal (i.e., 2, separate lesions in the same quadrant)/multi-centric (i.e., 2 separate lesions in different quadrants) tumors are allowed, as well as inflammatory breast cancer, and the tumor with the most advanced T stage should be used to assess the eligibility.
5. Provide a core needle biopsy consisting of at least 1 separate tumor-bearing cores from the primary tumor at screening for translational research (archival is acceptable if sufficient tumor is available; slides are acceptable if at least 15 are available)
6. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 assessed within 14 days of treatment initiation.
7. Demonstrate adequate organ function. All screening labs should be performed within 14 days of treatment initiation.
8. Have left ventricular ejection fraction (LVEF) of ≥50% or ≥ institution lower limit of normal (LLN) as assessed by echocardiogram (ECHO) or multigated acquisition (MUGA) scan performed at screening.
9. Males and female subjects of childbearing potential (Section 5.7.2 - Contraception) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 12 months after the last dose of study medication for subjects who have received cyclophosphamide, and 6 months after the last dose of study medication for subjects who did not.

   Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
10. (Female subject of childbearing potential) Have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or borderline a serum pregnancy test will be required.

Exclusion Criteria:

1. Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
2. Has received prior chemotherapy, targeted therapy, and radiation therapy within the past 12 months.
3. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) or has previously participated in MK-3475 clinical trials.
4. Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 4 weeks of the first dose of treatment in this current trial.

   Note: subject should be excluded if he/she received an investigational agent with anti-cancer or anti-proliferative intent within the last 12 months.
5. Has received a live vaccine within 30 days of the first dose of study treatment.

   Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines, and are not allowed.
6. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
7. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
8. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
9. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
10. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has significant cardiovascular disease, such as:

    * History of myocardial infarction, acute coronary syndrome or coronary angioplasty/stenting/bypass grafting within the last 6 months
    * Congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV or history of CHF NYHA class III or IV
13. Has a history or current evidence of any condition, therapy, lab abnormality or other circumstance that might expose the subject to risk by participating in the trial, confound the results of the trial, or interfere with the subject's participation for the full duration of the trial in the opinion of the Investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial in the opinion of the Investigator.
15. Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the screening visit through 12 months after the last dose of trial treatment for subjects who have received cyclophosphamide, and for 6 months after the last dose of study medication for subjects who have not.
16. Has a known hypersensitivity to the components of the study therapy or its analogs.
17. Has a known history of active TB (Bacillus Tuberculosis).
18. Allergy to ciprofloxacin (or other quinolones).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-07-08 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Arm A
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Arm A | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Customized [Median (Full Range); unit: years]
  Age, median | 56 [36 to 68] | 55 [31 to 66] | 55.5 [31 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12
Baseline ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) is a measure of functional status from scores ranging from 0 to 5. Baseline measure ECOG PS was collected during the screening physical exam.
  Participants
    ECOG PS 0 (Asymptomatic) | 6 | 6 | 12
    ECOG PS 1 (Symptomatic but completely ambulatory) | 0 | 0 | 0
    ECOG PS 2 (Symptomatic, <50% in bed during the day) | 0 | 0 | 0
    ECOG PS 3 (Symptomatic, >50% in bed, but not bedbound) | 0 | 0 | 0
    ECOG PS 4 (Bedbound) | 0 | 0 | 0
    ECOG PS 5 (Death) | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR) Rate (ypT0/Tis ypN0)
Description: Number of patients who showed pCR post surgery. pCR rate (ypT0/Tis ypN0) is defined as the proportion of subjects without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy per the current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery.
Time Frame: Following definitive surgery, approximately 9 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Arm A
Number analyzed (Participants) | 6 | 6
Participants | 2 | 5

2. Secondary Outcome: Safety and Tolerability Profile as Assessed by CTCAE v5.0
Description: Number of serious adverse events (SAE) reported by patients attributed to study drugs.
Time Frame: Cycle 1, Day 1 through safety follow-up visit, approximately 9 months.
Measure: Number; unit: Number of Occurrences
Arm/Group | Control | Arm A
Number analyzed (Participants) | 6 | 6
Number of Occurrences | 0 | 2

3. Secondary Outcome: Percent Change in Tumor Infiltrating Lymphocytes (TIL) Quantity Changes
Description: Evaluate increase in tumor infiltrating lymphocyte by H&E (comparing diagnostic biopsy to post-induction biopsy). Tumor infiltrating lymphocytes will be assessed by the San Antonio stromal TIL criteria.
Time Frame: Following definitive surgery, approximately 9 months.
Measure: Mean (95% Confidence Interval); unit: percentage change of TIL quantity
Arm/Group | Control | Arm A
Number analyzed (Participants) | 6 | 6
percentage change of TIL quantity | 11 [-36 to 59] | -26 [-58 to 5.6]

ADVERSE EVENTS:
Time Frame: From the start of study treatment through 90 days following the cessation of treatment or the initiation of new anti-cancer therapy (an average of 7 months).
Arm/Group | Control | Arm A
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=6) | Arm A (N=6)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=6) | Arm A (N=6)
Absolute neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 1 (1)
Bilateral leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 3 (5)
Injection site bruising (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Injection site erythema (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Lower leg tingling, intermittent (Nervous system disorders) | 1 (1) | 0 (0)
Mouth sores (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (4)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (5)
Peeling skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT04373031/Prot_SAP_000.pdf